CLINICAL TRIAL: NCT00079066
Title: A Phase III Randomized Study of Cetuximab (Erbitux™, C225) and Best Supportive Care Versus Best Supportive Care in Patients With Pretreated Metastatic Epidermal Growth Factor Receptor (EGFR)-Positive Colorectal Carcinoma
Brief Title: Cetuximab + Best Supportive Care Compared With Best Supportive Care Alone in Metastatic Epidermal Growth Factor Receptor-Positive Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Australasian Gastro-Intestinal Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO17; CAN-NCIC-CO17 (Other: PDQ); AGITG-CAN-NCIC-CO17 (Other: AGITG); BMS-CA225-025 (Other: Bristol-Myers Squibb); IMCL-CAN-NCIC-CO17 (Other: ImClone Systems Incorporated); CDR0000353486 (Other: PDQ)
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer; Quality of Life
Keywords: quality of life; stage IV colon cancer; recurrent colon cancer; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: cetuximab
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can target tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Best supportive care is the use of drugs and other treatments to improve the quality of life of patients. Combining cetuximab with best supportive care may slow the growth of the tumor and help patients live longer and more comfortably. It is not yet known whether cetuximab combined with best supportive care is more effective than best supportive care alone in treating metastatic epidermal growth factor receptor-positive colorectal cancer.

PURPOSE: This randomized phase III trial is studying cetuximab and best supportive care to see how well they work compared to best supportive care alone in treating patients with metastatic epidermal growth factor receptor-positive colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare survival of patients with metastatic epidermal growth factor receptor-positive colorectal cancer treated with cetuximab and best supportive care vs best supportive care alone.

Secondary

* Compare the time to disease progression in patients treated with these regimens.
* Compare the objective response rate in patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.
* Compare the health utilities of patients treated with these regimens.
* Conduct a comparative economic evaluation in patients treated with these regimens.
* Determine the safety profile of cetuximab in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to participating center and ECOG performance status (0 or 1 vs 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive an initial loading dose of cetuximab IV over 120 minutes on day 1. Patients continue to receive maintenance infusions of cetuximab IV over 60 minutes weekly. Patients also receive best supportive care, defined as measures designed to provide palliation of symptoms and improve quality of life as much as possible.
* Arm II: Patients receive best supportive care as in arm I. In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, and then at 4, 8, 16, and 24 weeks (or until deterioration to ECOG PS 4 or hospitalization for end-of-life care).

Patients are followed every 4 weeks.

PROJECTED ACCRUAL: A total of 500 patients (250 per treatment arm) will be accrued for this study within 20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer

  * Metastatic disease
* Epidermal growth factor receptor (EGFR)-positive by immunochemistry
* Measurable or evaluable disease
* Not amenable to standard curative therapy

  * Best supportive care is the only available option
* Must have received a prior thymidylate synthase inhibitor (e.g., fluorouracil, capecitabine, raltitrexed, or fluorouracil-uracil) in the adjuvant or metastatic setting

  * Combination therapy with oxaliplatin or irinotecan allowed
* Must have failed* a prior regimen containing irinotecan and a prior regimen containing oxaliplatin for metastatic disease OR relapsed within 6 months after an adjuvant regimen containing irinotecan or oxaliplatin OR have documented unsuitability for such regimens
* No symptomatic CNS metastases NOTE: *Failure is defined as either disease progression (clinical or radiological) or intolerance to the regimen

PATIENT CHARACTERISTICS:

Age

* 16 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics
* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 8.0 g/dL

Hepatic

* AST and ALT ≤ 5 times upper limit of normal (ULN)
* Bilirubin ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No uncontrolled angina
* No arrhythmias
* No cardiomyopathy
* No congestive heart failure
* No myocardial infarction* within the past 6 months NOTE: *Pre-treatment ECG as only evidence of infarction is allowed

Pulmonary

* No severe restrictive lung disease
* No interstitial lung disease by chest x-ray

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 4 weeks before, during, and for 4 weeks after study treatment
* No active pathological condition that would preclude study participation
* No psychological or geographical condition that would preclude study compliance
* No other malignancy within the past 5 years except adequately treated non-melanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior cetuximab
* No prior murine monoclonal antibody therapy (e.g., edrecolomab)

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy and recovered
* No concurrent chemotherapy

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* Concurrent palliative radiotherapy allowed except to index lesions

Surgery

* At least 4 weeks since prior major surgery and recovered

Other

* No prior EGFR-targeted therapy (e.g., erlotinib or gefitinib)
* More than 30 days since prior experimental therapeutic agents
* More than 4 weeks since prior investigational agents
* No concurrent enrollment in another clinical study
* No other concurrent EGFR-targeted therapy
* No other concurrent non-cytotoxic experimental agents

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2003-12-30 (Actual); Primary Completion 2006-11-03 (Actual); Study Completion 2009-02-10 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Time to progression
Objective response rate
Quality of life by European Organization for Research of the Treatment of Cancer Quality of Life Questionnaire -C30 (EORTC QLQ-C30)
Health utilities by Health Utilities Index 13 (HU 13)
Economic evaluation
Safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Derek Jonker, MD, Study Chair — Ottawa Regional Cancer Centre; Chris Karapetis, MD, Study Chair — National Health and Medical Research Council, Australia
Locations (33):
- NHMRC Clinical Trials Centre, Camperdown, New South Wales, Australia
- Canada (32):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Fraser Valley Cancer Centre at British Columbia Cancer Agency, Surrey, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre at Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Belleville General Hospital, Belleville, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Grand River Regional Cancer Centre at Grand River Hospital, Kitchener, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - R. S. McLaughlin Durham Regional Cancer Centre at Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Hotel Dieu Health Sciences Hospital - Niagara, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Care at Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto Sunnybrook Regional Cancer Centre at Sunnybrook and Women's College Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - St. Joseph's Health Centre - Toronto, Toronto, Ontario
  - Windsor Regional Cancer Centre at Windsor Regional Hospital, Windsor, Ontario
  - Prince Edward Island Cancer Centre at Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta A, O'Callaghan CJ, Zhu L, Jonker DJ, Wong RPW, Colwell B, Moore MJ, Karapetis CS, Tebbutt NC, Shapiro JD, Tu D, Booth CM. Evaluating the Time Toxicity of Cancer Treatment in the CCTG CO.17 Trial. JCO Oncol Pract. 2023 Jun;19(6):e859-e866. doi: 10.1200/OP.22.00737. Epub 2023 Mar 7. PMID 36881786
- [Result] Au HJ, Karapetis CS, O'Callaghan CJ, Tu D, Moore MJ, Zalcberg JR, Kennecke H, Shapiro JD, Koski S, Pavlakis N, Charpentier D, Wyld D, Jefford M, Knight GJ, Magoski NM, Brundage MD, Jonker DJ. Health-related quality of life in patients with advanced colorectal cancer treated with cetuximab: overall and KRAS-specific results of the NCIC CTG and AGITG CO.17 Trial. J Clin Oncol. 2009 Apr 10;27(11):1822-8. doi: 10.1200/JCO.2008.19.6048. Epub 2009 Mar 9. PMID 19273701
- [Result] Jonker DJ, Karapetis C, Harbison C, et al.: High epiregulin (EREG) gene expression plus K-ras wild-type (WT) status as predictors of cetuximab benefit in the treatment of advanced colorectal cancer (ACRC): results from NCIC CTG CO.17-A phase III trial of cetuximab versus best supportive care (BSC).. [Abstract] J Clin Oncol 27 (Suppl 15): A-4016, 2009.
- [Result] Asmis TR, Powell E, Karapetis CS, Jonker DJ, Tu D, Jeffery M, Pavlakis N, Gibbs P, Zhu L, Dueck DA, Whittom R, Langer C, O'Callaghan CJ. Comorbidity, age and overall survival in cetuximab-treated patients with advanced colorectal cancer (ACRC)--results from NCIC CTG CO.17: a phase III trial of cetuximab versus best supportive care. Ann Oncol. 2011 Jan;22(1):118-126. doi: 10.1093/annonc/mdq309. Epub 2010 Jul 5. PMID 20603436
- [Result] Karapetis CS, Khambata-Ford S, Jonker DJ, O'Callaghan CJ, Tu D, Tebbutt NC, Simes RJ, Chalchal H, Shapiro JD, Robitaille S, Price TJ, Shepherd L, Au HJ, Langer C, Moore MJ, Zalcberg JR. K-ras mutations and benefit from cetuximab in advanced colorectal cancer. N Engl J Med. 2008 Oct 23;359(17):1757-65. doi: 10.1056/NEJMoa0804385. PMID 18946061
- [Result] Mittmann N, Au HJ, Tu D, et al.: A prospective economic analysis of cost-effectiveness of cetuximab for metastatic colorectal cancer patients from the NCIC CTG and AGITG CO.17 trial. [Abstract] J Clin Oncol 26 (Suppl 15): A-6528, 2008.
- [Result] O'Callaghan CJ, Tu D, Karapetis CS, et al.: The relationship between the development of rash and clinical and quality of life outcomes in colorectal cancer patients treated with cetuximab in NCIC CTG CO.17. [Abstract] J Clin Oncol 26 (Suppl 15): A-4130, 2008.
- [Result] Jonker DJ, Karapetis CS, Moore M, et al.: Randomized phase III trial of cetuximab monotherapy plus best supportive care (BSC) versus BSC alone in patients with pretreated metastatic epidermal growth factor receptor (EGFR)-positive colorectal carcinoma: a trial of the National Cancer Institute of Canada Clinical Trials Group (NCIC CTG) and the Australasian Gastro-Intestinal Trials Group (AGITG). [Abstract] American Association for Cancer Research: 98th Annual Meeting, April 14-18, 2007, Los Angeles, CA. 2007.
- [Result] Jonker DJ, O'Callaghan CJ, Karapetis CS, Zalcberg JR, Tu D, Au HJ, Berry SR, Krahn M, Price T, Simes RJ, Tebbutt NC, van Hazel G, Wierzbicki R, Langer C, Moore MJ. Cetuximab for the treatment of colorectal cancer. N Engl J Med. 2007 Nov 15;357(20):2040-8. doi: 10.1056/NEJMoa071834. PMID 18003960
- [Derived] Nicholls DL, Xu MC, Zhan L, Sharma D, Hueniken K, Chiasson K, Wahba M, Brown MC, Grant B, Shapiro J, Karapetis CS, Simes J, Jonker D, Tu D, O'Callaghan C, Chen E, Liu G. Machine Learning Models of Early Longitudinal Toxicity Trajectories Predict Cetuximab Concentration and Metastatic Colorectal Cancer Survival in the Canadian Cancer Trials Group/AGITG CO.17/20 Trials. JCO Clin Cancer Inform. 2025 Apr;9:e2400114. doi: 10.1200/CCI.24.00114. Epub 2025 Apr 11. PMID 40215447
- [Derived] Gupta A, O'Callaghan CJ, Zhu L, Jonker DJ, Wong RPW, Colwell B, Moore MJ, Karapetis CS, Tebbutt NC, Shapiro JD, Tu D, Booth CM. The association of health-care contact days with physical function and survival in CCTG/AGITG CO.17. J Natl Cancer Inst. 2024 Aug 1;116(8):1313-1318. doi: 10.1093/jnci/djae077. PMID 38656931
- [Derived] Loree JM, Dowers A, Tu D, Jonker DJ, Edelstein DL, Quinn H, Holtrup F, Price T, Zalcberg JR, Moore MJ, Karapetis CS, O'Callaghan CJ, Waring P, Kennecke HF, Hamilton SR, Kopetz S. Expanded Low Allele Frequency RAS and BRAF V600E Testing in Metastatic Colorectal Cancer as Predictive Biomarkers for Cetuximab in the Randomized CO.17 Trial. Clin Cancer Res. 2021 Jan 1;27(1):52-59. doi: 10.1158/1078-0432.CCR-20-2710. Epub 2020 Oct 21. PMID 33087330
- [Derived] Hay AE, Pater JL, Corn E, Han L, Camacho X, O'Callaghan C, Chong N, Bell EN, Tu D, Earle CC. Pilot study of the ability to probabilistically link clinical trial patients to administrative data and determine long-term outcomes. Clin Trials. 2019 Feb;16(1):14-17. doi: 10.1177/1740774518815653. Epub 2018 Nov 22. PMID 30466310